CLINICAL TRIAL: NCT01657292
Title: Open, Blindly Evaluated, Prospective, Controlled, Randomized, Multicenter Phase III Clinical Trial to Compare Intra-individually the Efficacy and Tolerance of Oleogel-S10 Versus Standard of Care in Accelerating the Healing of Grade 2a Partial-Thickness Burn Wounds
Brief Title: Oleogel-S10 Versus Standard of Care in Healing of Grade 2a Burn Wounds
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Birken AG (Industry)
Responsible Party: Sponsor
Organization: Amryt Pharma (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BBW-11; 2012-000362-38 (EudraCT Number)
Record Dates: First submitted 2012-07-29; First posted 2012-08-06 (Estimated); Results first posted 2015-09-28 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-08

CONDITIONS: Burns
Keywords: Wound healing; Burn wound; Superficial partial-thickness burn wound; Grade 2a burn wounds; Time to wound closure
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oleogel-S10 ointment (Experimental): Intra-individual comparison. Oleogel-S10 ointment is administered to one randomly assigned wound half.
  Interventions: Drug: Oleogel-S10 ointment; Device: Octenilin® wound gel
- Octenilin® wound gel (Other): Intraindividual comparison: The other wound half receives disinfectant Octenilin® wound gel.
  Interventions: Drug: Oleogel-S10 ointment; Device: Octenilin® wound gel

INTERVENTIONS:
Drug: Oleogel-S10 ointment — Intraindividual comparison: One randomly assigned wound half is treated with Oleogel-S10 ointment and fatty gauze wound dressing
Device: Octenilin® wound gel — Intraindividual comparison: The other wound half is treated with Octenilin® wound gel and fatty gauze wound dressing
  Other Names: Contains Octenidine

SUMMARY:
The main goal of this phase III clinical trial is to show safety and efficacy of Oleogel-S10 in the acceleration of wound healing of grade 2a burn wounds.

DETAILED DESCRIPTION:
Oleogel-S10 has shown efficacy and was well tolerated in previous clinical trials in patients with skin lesions. Especially the results in the split-thickness skin graft donor site, which is regarded as an excellent model for any kind of superficial wounds in human skin, suggest that Oleogel-S10 should be efficacious and safe in treatment of grade 2a burns.

The present Phase III clinical trial in grade 2a burns is initiated in order to measure the wound healing progress applying objective methods, i.e., the time to healing and the grade of epithelialization of the wound.

In this study, grade 2a burn wounds are separated into two halves: Following wound cleaning and disinfection, wounds are separated into two wound halves. Randomly assigned, one wound half receives Oleogel-S10 ointment, the other wound half standard of care treatment.

Wound healing progress is documented by photos which are assessed by expert reviewers blinded to the treatment of the wound halves.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years old who have provided written informed consent.
* Presenting with acute grade 2a burn wounds (as graded by an expert surgeon assisted by LDI or a multispectral imaging system) within 48 hours after injury.
* Burn wound caused by fire burn, heat burn or scalding.
* Burn patients with grade 2a burn wounds between 80 cm2 and less than 25% of their TBSA (alternatively, 2 comparable wounds with size more than 40 cm2 each and less than 12.5% of the TBSA each are allowed).
* Patient is able to understand the Informed Consent Form provided and is prepared to comply with all study requirements, including the following: Visiting the trial site for wound dressing changes at least every second day (if patient is not hospitalized) and photo documentation until full wound closure or until the Investigator decides to change medication and/or treatment after day 21 after start of treatment
* Willing to perform all necessary wound dressing changes at the trial site. Also the patient needs to agree to return to site for 3 and 12 months follow-up visits.
* Women of childbearing potential must apply highly effective method of birth control (failure rate less than 1% per year when used consistently and correctly (e.g., implants, injectables, combined oral contraceptives, some intrauterine contraceptive devices (IUDs), sexual abstinence, or a vasectomized partner))

Exclusion Criteria:

* Suffering from chemical burns, or electrical burns or sunburns
* Having already received treatment for their burn with silver sulfadiazine (obscures photographic wound evaluation).
* Positive blood culture after the burn.
* Diseases or conditions that could, in the opinion of the Investigator, interfere with the assessment of safety, tolerance or efficacy.
* A skin disorder that is chronic or currently active and which the Investigator considers will adversely affect the healing of the acute wounds or involves the areas to be examined in this trial.
* A history of clinically significant hypersensitivity to any of the drugs or surgical dressings to be used in this trial.
* Known multiple allergic disorders.
* Taking, or have taken, any investigational drugs within 3 months prior to the screening visit.
* Pregnant or breast feeding women are not allowed to participate in the study.
* Inappropriate to participate in the study, for any reason, in the opinion of the Investigator.
* Mental incapacity or language barriers precluding adequate understanding or co-operation or willingness to follow study procedures.
* Previous participation in this study.
* Employee at the investigational site, relative or spouse of the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2012-08; Primary Completion 2013-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Hartmann, Dr., Principal Investigator — Trauma Hospital Berlin, Warener Str. 7, 12683 Berlin, Germany
Locations (9):
- Germany (3):
  - Unfallkrankenhaus Berlin, Berlin
  - Berufsgenossenschaftliches Universitätsklinikum Bergmannsheil, Bochum
  - Universitätsklinikum Schleswig-Holstein, Lübeck
- Sweden (2):
  - Linköping University Hospital, Linköping
  - University Hospital, Uppsala
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland
- United Kingdom (3):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Broomfield Hospital, Chelmsford
  - Queen Victoria Hospital, East Grinstead

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 31-Aug-2012 to 10-Jul-2013, in 10 clinical centres in 4 countries: Germany (4 centers), Uk (3 centers), Sweden (2 centers), and Switzerland (1 center).
Pre-assignment Details: 66 patients were screened of which 5 violated eligibility criteria and thus 61 subjects were treated.
Groups:
- Entire Study Population: All patients treated with Oleogel-S10 and Octenilin® wound gel.
Period: Overall Study
Arm/Group | Entire Study Population
Started | 61
Completed | 51
Not Completed | 10
Not completed — Adverse Event | 6
Not completed — Withdrawal by Subject | 2
Not completed — Violation of eligibility criteria | 1
Not completed — Change of therapy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Entire Study Population
Number analyzed (Participants) | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 54
  >=65 years | 6
Age, Continuous [Median (Full Range); unit: years] | 41 [18 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 42
Region of Enrollment [Number; unit: participants]
  Sweden | 3
  United Kingdom | 28
  Switzerland | 4
  Germany | 26

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Earlier Healing of the Wound Half Treated With Oleogel-S10 Compared to the Wound Half Receiving Standard of Care
Description: Photo-based evaluation by independent experts blinded to the treatment regime.
Time Frame: 2 to 3 weeks
Population: The analysis included all patients who were treated at least once with Oleogel-S10 or Octenilin® wound gel (as randomised) and for whom a difference in wound healing between the treatment was observed.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Entire Study Population
Number analyzed (Participants) | 35
percentage of patients | 85.7 [69.7 to 95.2]
Statistical Analysis 1: Comparison: Entire Study Population; All patients received both treatments and treatments were intra-individually compared. Hypotheses tested: H0: s0 ≤0.5 and H1: s0 >0.5 (with s0=rate of superiority of Oleogel-S10); Test type: Superiority or Other; p < 0.0001, Binomial test — 1-sided, significance level = 0.025

2. Secondary Outcome: Intra-individual Difference in Time to Wound Closure Between Wound Halves, Either Treated With Oleogel-S10 or Treated With Standard of Care
Time Frame: 2 to 3 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Time From Study Start After Burn Accident Until Wound Closure is Achieved Separately for Wound Halves Treated With Oleogel-S10 vs. Standard of Care
Time Frame: 2 to 3 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Percentage of Patients With Wound Closure at Different Time Points
Time Frame: 2 to 3 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Percentage of Wound Epithelialization at Different Time Points as Assessed by the Investigator
Time Frame: 2 to 3 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Likert Scale Rating of Efficacy (Evaluated by Both the Investigators and Patients)
Description: By direct comparison of the separate simultaneous treatments for the two wound halves, patients and investigators, respectively, are asked to grade the efficacy of Oleogel-S10 Versus Standard of Care on a questionnaire with a 5-point graded visual analogue scale
Time Frame: 2 to 3 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Cosmetic Outcome After 3 and 12 Months After Burn Accident, in Relation to Texture, Redness, Growth of Hair and Pigmentation, Based on Blinded Photo Evaluation
Time Frame: 3 and 12 months
Reporting Status: Not Posted

8. Secondary Outcome: Likert Scale Rating of Tolerance (Evaluated by Both the Investigators and Patients)
Description: By direct comparison of the separate simultaneous treatments for the two wound halves, patients and investigators, respectively, are asked to provide their opinion on the tolerance of Oleogel-S10 Versus Standard of Care on a questionnaire with a 5-point graded visual analogue scale
Time Frame: 2 to 3 weeks
Reporting Status: Not Posted

9. Secondary Outcome: PK Data: Systemic Presence/Concentration of Betulin in Blood Plasma Samples
Time Frame: 2 to 3 weeks
Reporting Status: Not Posted

10. Secondary Outcome: Microbial Colonization of the Wound Halves
Time Frame: 2 to 3 weeks
Reporting Status: Not Posted

11. Secondary Outcome: Assessment of Adverse Events
Time Frame: 2 to 3 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Day 0 (start of treatment) till end of treatment (Day 21 or earlier if full wound closure was achieved earlier, or later, if the investigator decided to change medication and/or treatment due to unsatisfying wound closure after Day 21).
Groups:
- Entire Study Population - Systemic AEs: All patients treated with Oleogel-S10 and Octenilin® wound gel. Systemic AEs which are not localized to the wound application site are reported under this arm.
- Oleogel-S10 Localized AE: All patients treated with Oleogel-S10 and Octenilin® wound gel. Application site reactions which occurred only at the Oleogel-S10 wound half are reported under this arm.
- Octenilin Localized AE: All patients treated with Oleogel-S10 and Octenilin® wound gel. Application site reactions which occurred only at the Octenilin® wound half are reported under this arm.
- Localized AE Both Wound Halves: All patients treated with Oleogel-S10 and Octenilin® wound gel. Application site reactions which occurred at both the Octenilin® wound half and Oleogel-S10 wound half in one patient are reported under this arm.
Arm/Group | Entire Study Population - Systemic AEs | Oleogel-S10 Localized AE | Octenilin Localized AE | Localized AE Both Wound Halves
Serious Adverse Events (participants affected / at risk) | 2/61 | 1/61 | 1/61 | 4/61
Other Adverse Events (participants affected / at risk) | 0/61 | 0/61 | 0/61 | 0/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Entire Study Population - Systemic AEs (N=61) | Oleogel-S10 Localized AE (N=61) | Octenilin Localized AE (N=61) | Localized AE Both Wound Halves (N=61)
Wound necrosis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Condition aggravated (General disorders) | 0 | 0 | 0 | 2 — Further deepening of burn wound
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication requires approval of the sponsor without specification of an embargo time period.